CLINICAL TRIAL: NCT06516770
Title: The Effects of Different Types of Stimulation on Movement Control and Motor Unit Behavior in Individuals With Lumbopelvic Movement Control Impairment
Brief Title: Movement Control and Motor Unit Behavior Responses to Different Types of Stimulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Peemongkon Wattananon, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-CIRB 2022/118.0711
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain
Keywords: Transcranial direct current stimulation; Neuromuscular electrical stimulation; Motor control exercise; Isometric exercise; Motor unit behavior; Movement control; Lumbar multifidus muscle
MeSH Terms: conditions — Low Back Pain | interventions — Transcranial Direct Current Stimulation; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transcranial direct current stimulation (Experimental): The subject will receive transcranial direct current stimulation for 20 minutes.
  Interventions: Device: Transcranial direct current stimulation
- Neuromuscular electrical stimulation (Experimental): The subject will receive neuromuscular electrical stimulation for 20 minutes.
  Interventions: Device: Neuromuscular electrical stimulation
- Motor control exercise (Experimental): The subject will receive motor control exercise for 20 minutes.
  Interventions: Other: Motor control exercise
- Isometric exercise (Active Comparator): The subject will receive isometric exercise for 20 minutes.
  Interventions: Other: Isometric exercise

INTERVENTIONS:
Device: Transcranial direct current stimulation — The subject will receive the tDCS using 5X7 cm electrodes. The anodal electrode will be placed on M1 representing the back muscles (1 cm anterior and 4 cm lateral to the vertex), while cathodal electrode will be placed on contralateral supraorbital area. The intensity will be set at 2 mA with 10-second fade in/out. The subject will be stimulated by tDCS for 20 minutes
  Arms: Transcranial direct current stimulation
Device: Neuromuscular electrical stimulation — The participants will receive the NMES using interferential mode (6000 Hz, beat frequency 20-50 Hz, scanning effect) on bilateral LM. The intensity will be set at the subject's maximum tolerance. Stimulation will be set at 10 seconds on and 60 seconds off to minimize muscle fatigue. The total NMES time is 20 minutes.
  Arms: Neuromuscular electrical stimulation
Other: Motor control exercise — The participant will be instructed to perform co-contraction of transverse abdominis and lumbar multifidus muscle, while performing self-selected pace forward bend. Emphasis will be given to move in control manner (smooth and symmetrical movement). The participant will perform 4 minutes of continuous movement for 4 sets with 1 minute rest between sets.
  Arms: Motor control exercise
Other: Isometric exercise — The participant will be instructed to perform isometric back extension exercise in modified Sorensen position. The participant will hold 60 seconds in neutral position for 5 repetitions with 3 minutes rest between repetitions.
  Arms: Isometric exercise

SUMMARY:
This study aims to determine the effect of different stimulations including 1) transcranial direct current stimulation (tDCS), 2) neuromuscular electrical stimulation (NMES), 3) motor control exercise (MCE), and 4) isometric exercise (IE) on movement control and motor unit behavior in individuals with movement control impairment, and determine the correlation between movement control and motor unit behavior.

DETAILED DESCRIPTION:
After obtaining the written informed consent, all participants will fill out the information sheet for demographic data. Data collection will be conducted in private laboratory with closed environment. Only lab staffs can access to the lab. Female researchers will perform participant preparation. Participants will be informed that they have to change their cloth to lab tank top to expose their lower back area. However, they can decline to change their cloth. In this case, researchers will fold their cloth to expose the lower back. The body landmarks will be identified. These landmarks include 1) spinous processes (L1 and S1 levels), 2) lumbar multifidus (LM) (2 cm lateral to lower half of L4 spinous process), 3) bilateral lateral epicondyle of femur, and 4) bilateral lateral malleolus. Spinous process of L1, S2, bilateral lateral epicondyle of femur, and bilateral lateral malleolus will be used as locations for inertial measurement unit (IMU) sensors, while LM location will be used to place surface electrode for decomposition electromyography (dEMG). This preparation process will take about 20 minutes.

The participant will be asked to perform 1-minute active forward bend based on speed and load that can differentiate between healthy individuals and individuals with movement control impairment. IMU and dEMG data are concurrently collected. Five-minute rest will be provided to avoid muscle fatigue. After that, participant will be randomly assigned to one of four stimulations including transcranial direct current stimulation (tDCS), neuromuscular electrical stimulation (NMES), isometric exercise (IE), and motor control exercise (MCE). Each stimulation will take approximately 20 minutes.

Types of stimulation Transcranial direct current stimulation (tDCS): The participant will receive the tDCS using 5X7 cm electrodes. The anodal electrode will be placed on M1 representing the back muscles (1 cm anterior and 4 cm lateral to the vertex), while cathodal electrode will be placed on contralateral supraorbital area. The intensity will be set at 2 mA with 10-second fade in/out. The subject will be stimulated by tDCS for 20 minutes.

Neuromuscular electrical stimulation (NMES): The participants will receive the NMES using interferential mode (6000 Hz, beat frequency 20-50 Hz, scanning effect) on bilateral LM. The intensity will be set at the subject's maximum tolerance. Stimulation will be set at 10 seconds on and 60 seconds off to minimize muscle fatigue. The total NMES time is 20 minutes.

Isometric exercise (IE): The participant will be instructed to perform isometric back extension exercise in modified Sorensen position. The participant will hold 60 seconds in neutral position for 5 repetitions with 3 minutes rest between repetitions.

Movement control exercise (MCE): The participant will be instructed to perform co-contraction of transverse abdominis and lumbar multifidus muscle, while performing self-selected pace forward bend. Emphasis will be given to move in control manner (smooth and symmetrical movement). The participant will perform 4 minutes of continuous movement for 4 sets with 1 minute rest between sets. This exercise is low intensity focusing on control of movement; therefore, the occurrence of muscle fatigue is unlikely.

After completion of one session stimulation, the participant will be asked to perform 1-minute active forward bend with the same speed and load again, while IMU and dEMG data will be simultaneously corrected. IMU data will be used to determine the effect of stimulation (tDCS, NMES, IE, and MCE) on movement control in individuals with movement control impairment. dEMG data will be used to determine the effect of each stimulation on motor unit behavior (spatial and temporal motor unit recruitment). In addition, IMU and dEMG data will be further used to determine the association between movement control and motor unit behavior. Data collection including 20-minute stimulation will take approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 40
2. Both male and female
3. Presence of movement control impairment (instability catch during clinical observation of active forward bend test)
4. No current episode of low back pain
5. No definitive neurologic signs including weakness or numbness in the lower extremity
6. No previous spinal surgery
7. Have not been diagnosed osteoporosis, severe spinal stenosis, inflammatory joint disease, and/or systemic disease
8. Body mass index (BMI) less than 30 kg/m2

Exclusion Criteria:

1. Pregnancy
2. Any lower extremity condition that would potentially alter trunk movement in standing
3. Vestibular dysfunction
4. Extreme psychosocial involvement
5. Active treatment of another medical illness that would preclude participation in any aspect of the study
6. Contraindication for tDCS including a history of head injury/surgery, seizure, cardiac pacemaker, metal/electrical/magnetic implantation, uncontrolled migraine headache

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Segmental angular velocity in degrees/second | baseline and immediately after the intervention
  Segmental angular velocity will be derived from the inertial measurement units.
Clinical observation | baseline and immediately after the intervention
  Clinical observation rating will be recorded as presence or absence of aberrant movement by two raters.
Number of motor units | baseline and immediately after the intervention
  Number of motor units will be derived from decomposition of muscle activity using electromyography system.
Motor unit action potential in millivolts | baseline and immediately after the intervention
  Motor unit action potential will be derived from decomposition of muscle activity using electromyography system.
Motor unit firing rate in pulses/second | baseline and immediately after the intervention
  Motor unit firing rate will be derived from decomposition of muscle activity using electromyography system.

SECONDARY OUTCOMES:
Pain intensity | baseline
  Pain intensity will be evaluated using numeric pain rating scale. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine" or "worst pain imaginable".
Level of disability in percentage | baseline
  Level of disability will be evaluated using modified Oswestry Disability Questionnaire. Questionnaire examines the level of disability in 10 everyday activities of daily living. Each item consist of 6 statements which are scored from 0 to 5. With 0 indicating the least disability and 5 the greatest then the total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability.
Fear of movement level | baseline
  Fear of movement will be evaluated using Tampa Scale for Kinesiophobia. The 17-item Tampa Scale for Kinesiophobia total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Perception of change | immediately after the intervention
  Perception of change will be evaluated using a Global Rating of Change Questionnaire. It is composed of a scale (-4 to +4) that assesses whether the patient condition has gotten worse, better, or stayed the same and to quantify the magnitude of that change after exercise. In the middle of the response scale is a "0" indicating no improvement or no change, the negative values towards the left indicate worsening symptoms or a deterioration in status, and positive values towards the right indicate improvement in the health status.

CONTACTS AND LOCATIONS:
Overall Officials: Peemongkon Wattananon, PhD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

REFERENCES:
- [Background] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Background] O'Sullivan P. Diagnosis and classification of chronic low back pain disorders: maladaptive movement and motor control impairments as underlying mechanism. Man Ther. 2005 Nov;10(4):242-55. doi: 10.1016/j.math.2005.07.001. Epub 2005 Sep 9. PMID 16154380
- [Background] Sahrmann S, Azevedo DC, Dillen LV. Diagnosis and treatment of movement system impairment syndromes. Braz J Phys Ther. 2017 Nov-Dec;21(6):391-399. doi: 10.1016/j.bjpt.2017.08.001. Epub 2017 Sep 27. PMID 29097026
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377
- [Background] Panjabi MM. Clinical spinal instability and low back pain. J Electromyogr Kinesiol. 2003 Aug;13(4):371-9. doi: 10.1016/s1050-6411(03)00044-0. PMID 12832167
- [Background] Reeves NP, Cholewicki J, van Dieen JH, Kawchuk G, Hodges PW. Are Stability and Instability Relevant Concepts for Back Pain? J Orthop Sports Phys Ther. 2019 Jun;49(6):415-424. doi: 10.2519/jospt.2019.8144. Epub 2019 Apr 25. PMID 31021689
- [Background] van Dieen JH, Reeves NP, Kawchuk G, van Dillen LR, Hodges PW. Motor Control Changes in Low Back Pain: Divergence in Presentations and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):370-379. doi: 10.2519/jospt.2019.7917. Epub 2018 Jun 12. PMID 29895230
- [Background] Biely SA, Silfies SP, Smith SS, Hicks GE. Clinical observation of standing trunk movements: what do the aberrant movement patterns tell us? J Orthop Sports Phys Ther. 2014 Apr;44(4):262-72. doi: 10.2519/jospt.2014.4988. Epub 2014 Jan 22. PMID 24450372
- [Background] Kong-Oun S, Prasertkul W, Fungkiatphaiboon P, Wattananon P. The inter-rater reliability of clinical observation of prone hip extension and association between aberrant movement and chronic low back pain. Musculoskelet Sci Pract. 2022 Feb;57:102476. doi: 10.1016/j.msksp.2021.102476. Epub 2021 Nov 6. PMID 34768224
- [Background] Luomajoki H, Kool J, de Bruin ED, Airaksinen O. Movement control tests of the low back; evaluation of the difference between patients with low back pain and healthy controls. BMC Musculoskelet Disord. 2008 Dec 24;9:170. doi: 10.1186/1471-2474-9-170. PMID 19108735
- [Background] Wattananon P, Ebaugh D, Biely SA, Smith SS, Hicks GE, Silfies SP. Kinematic characterization of clinically observed aberrant movement patterns in patients with non-specific low back pain: a cross-sectional study. BMC Musculoskelet Disord. 2017 Nov 15;18(1):455. doi: 10.1186/s12891-017-1820-x. PMID 29141615
- [Background] Laird RA, Kent P, Keating JL. Modifying patterns of movement in people with low back pain -does it help? A systematic review. BMC Musculoskelet Disord. 2012 Sep 7;13:169. doi: 10.1186/1471-2474-13-169. PMID 22958597
- [Background] Khobkhun F, Hollands MA, Richards J, Ajjimaporn A. Can We Accurately Measure Axial Segment Coordination during Turning Using Inertial Measurement Units (IMUs)? Sensors (Basel). 2020 Apr 29;20(9):2518. doi: 10.3390/s20092518. PMID 32365573
- [Background] Seel T, Raisch J, Schauer T. IMU-based joint angle measurement for gait analysis. Sensors (Basel). 2014 Apr 16;14(4):6891-909. doi: 10.3390/s140406891. PMID 24743160
- [Background] Hodges PW, Coppieters MW, MacDonald D, Cholewicki J. New insight into motor adaptation to pain revealed by a combination of modelling and empirical approaches. Eur J Pain. 2013 Sep;17(8):1138-46. doi: 10.1002/j.1532-2149.2013.00286.x. Epub 2013 Jan 25. PMID 23349066
- [Background] Wattananon P, Silfies SP, Tretriluxana J, Jalayondeja W. Lumbar Multifidus and Erector Spinae Muscle Synergies in Patients with Nonspecific Low Back Pain During Prone Hip Extension: A Cross-sectional Study. PM R. 2019 Jul;11(7):694-702. doi: 10.1002/pmrj.12002. Epub 2019 Feb 27. PMID 30811878
- [Background] Wattananon P, Sinsurin K, Somprasong S. Association between lumbopelvic motion and muscle activation in patients with non-specific low back pain during forward bending task: A cross-sectional study. Hong Kong Physiother J. 2020 Jun;40(1):29-37. doi: 10.1142/S1013702520500043. Epub 2019 Dec 30. PMID 32489238
- [Background] De Luca CJ. Control properties of motor units. J Exp Biol. 1985 Mar;115:125-36. doi: 10.1242/jeb.115.1.125. PMID 4031760
- [Background] De Luca CJ, Contessa P. Biomechanical benefits of the Onion-Skin motor unit control scheme. J Biomech. 2015 Jan 21;48(2):195-203. doi: 10.1016/j.jbiomech.2014.12.003. Epub 2014 Dec 9. PMID 25527890
- [Background] Merletti R, Knaflitz M, DeLuca CJ. Electrically evoked myoelectric signals. Crit Rev Biomed Eng. 1992;19(4):293-340. PMID 1563271
- [Background] De Luca CJ, Chang SS, Roy SH, Kline JC, Nawab SH. Decomposition of surface EMG signals from cyclic dynamic contractions. J Neurophysiol. 2015 Mar 15;113(6):1941-51. doi: 10.1152/jn.00555.2014. Epub 2014 Dec 24. PMID 25540220
- [Background] Nawab SH, Chang SS, De Luca CJ. High-yield decomposition of surface EMG signals. Clin Neurophysiol. 2010 Oct;121(10):1602-15. doi: 10.1016/j.clinph.2009.11.092. Epub 2010 Apr 28. PMID 20430694
- [Background] Silva MF, Dias JM, Pereira LM, Mazuquin BF, Lindley S, Richards J, Cardoso JR. Determination of the motor unit behavior of lumbar erector spinae muscles through surface EMG decomposition technology in healthy female subjects. Muscle Nerve. 2017 Jan;55(1):28-34. doi: 10.1002/mus.25184. Epub 2016 Nov 1. PMID 27170098
- [Background] Doucet BM, Lam A, Griffin L. Neuromuscular electrical stimulation for skeletal muscle function. Yale J Biol Med. 2012 Jun;85(2):201-15. Epub 2012 Jun 25. PMID 22737049
- [Background] Mariano TY, Burgess FW, Bowker M, Kirschner J, Van't Wout-Frank M, Jones RN, Halladay CW, Stein M, Greenberg BD. Transcranial Direct Current Stimulation for Affective Symptoms and Functioning in Chronic Low Back Pain: A Pilot Double-Blinded, Randomized, Placebo-Controlled Trial. Pain Med. 2019 Jun 1;20(6):1166-1177. doi: 10.1093/pm/pny188. PMID 30358864
- [Background] Nussbaum EL, Houghton P, Anthony J, Rennie S, Shay BL, Hoens AM. Neuromuscular Electrical Stimulation for Treatment of Muscle Impairment: Critical Review and Recommendations for Clinical Practice. Physiother Can. 2017;69(5):1-76. doi: 10.3138/ptc.2015-88. PMID 29162949
- [Background] Songjaroen S, Sungnak P, Piriyaprasarth P, Wang HK, Laskin JJ, Wattananon P. Combined neuromuscular electrical stimulation with motor control exercise can improve lumbar multifidus activation in individuals with recurrent low back pain. Sci Rep. 2021 Jul 20;11(1):14815. doi: 10.1038/s41598-021-94402-2. PMID 34285318
- [Background] Schabrun SM, Jones E, Elgueta Cancino EL, Hodges PW. Targeting chronic recurrent low back pain from the top-down and the bottom-up: a combined transcranial direct current stimulation and peripheral electrical stimulation intervention. Brain Stimul. 2014 May-Jun;7(3):451-9. doi: 10.1016/j.brs.2014.01.058. Epub 2014 Jan 30. PMID 24582372
- [Background] Aasa B, Berglund L, Michaelson P, Aasa U. Individualized low-load motor control exercises and education versus a high-load lifting exercise and education to improve activity, pain intensity, and physical performance in patients with low back pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2015 Feb;45(2):77-85, B1-4. doi: 10.2519/jospt.2015.5021. PMID 25641309